CLINICAL TRIAL: NCT07229677
Title: The AEVI-Fiji Cohort Study: a Longitudinal Study Assessing the Transmission Risk and Dynamics of Mosquito-borne and Respiratory Viruses in Fiji.
Brief Title: Cohort Study of Arbovirus and Other Emerging Virus Infections in Fiji: AEVI-Fiji Cohort.
Acronym: AEVI-Fiji
Status: Recruiting | Type: Observational
Sponsor: Fiji National University (Other)
Collaborators: Institut Louis Malardé (Other); Institut Pasteur (Industry); Institut Hospitalo-Universitaire Méditerranée Infection (Other); Ministry of Health, Fiji (Other Government); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: FNUHHREC 017.25; FNHRERC 08/25 (Other: Fiji National Health Research Ethics Review Committee)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Arbovirus Infections; Respiratory Infection Virus
Keywords: Seroprevalence; Longitudinal cohort; Respiratory viruses; Arboviruses; Fiji Islands
MeSH Terms: conditions — Arbovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected by trained phlebotomists at each scheduled visit (V1 to V4) as follows:
  * Participants aged 12 years and older: whole blood will be collected; serum will be extracted and stored at -80°C.
  * Participants aged 6-11 years: capillary blood will be collected on filter paper, dried, and stored at -4°C.
  Each participant will be assigned a unique Participant ID to ensure pseudonymization. The ID consists of a 4-digit participant number combined with a 7-character visit code (e.g., AEVI-FV1 to AEVI-FV4) to differentiate study visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Households members representative of the Fijian population (6 years and older): The study sample comprises randomly selected households from 30 Enumeration Areas (EAs) within the Central Division, selected in proportion to population size to ensure representativeness of the Fijian population. Both urban and rural settings are included. All individuals aged 6 years and above residing for more than 6 months in the selected households are invited to participate in the study.

SUMMARY:
Background: Fiji, an archipelago in the South Pacific comprising 332 islands distributed among 4 health administrative divisions (Central, Western, Eastern, Northern), is particularly vulnerable to the (re-)emergence of arboviruses and respiratory viruses due to its sub-tropical climate, the presence of several mosquito vector species, and connections with many countries in the Pacific, Asia and North America. Over the past decades, the epidemiological landscape of arboviruses has shifted from the sequential circulation of each of the four dengue virus (DENV) serotypes to the emergence of Zika virus (ZIKV) and chikungunya virus (CHIKV), concomitantly to the concurrent circulation of multiple DENV serotypes. The emergence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in 2020 significantly challenged Fiji's healthcare system, with the Delta variant alone accounting for approximately 700 deaths, while other respiratory viruses, such as influenza A and B, cause seasonal outbreaks. Despite these threats, comprehensive and up-to-date seroprevalence data remain scarce, limiting the capacity to inform and adapt public health policies.

Methods: The cohort study of Arbovirus and other Emerging Virus Infections in Fiji (AEVI-Fiji cohort study) aims to estimate the prevalence of several arboviruses and respiratory viruses, track the evolution of individual immunity, and analyse transmission dynamics of these viruses within the Fijian population. This longitudinal study will span 38 months and will include about 900 willing participants aged six years and older, recruited from at least 210 households randomly selected across the Central Division. Four visits will be conducted 12 months apart in each household. During each visit, participants will complete a questionnaire capturing their demographic characteristics and history of infections with major arboviruses and respiratory viruses and will provide a blood sample for serological analysis. During the whole study period, participants with a suspected acute infection by an arbovirus or respiratory virus will be screened.

Discussion: For the first time in Fiji, the AEVI-Fiji cohort study will generate longitudinal data to explore the determinants of both arbovirus and respiratory virus infections. The findings are expected to guide targeted public health strategies and enhance preparedness for future infectious disease threats in Fiji and the broader Oceania region.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 6 years and older who reside in the Central Division of Fiji
* Have lived in the selected household for at least six months at the time of enrollment

Exclusion Criteria:

* Pregnant women;
* Women in labor, or breastfeeding mothers;
* Individuals deprived of liberty by judicial or administrative decision;
* Individuals under psychiatric care or admitted to a health or social care facility for purposes other than participation in the study;
* Adults under legal protection or unable to provide informed consent;
* Homeless individuals;
* Individuals with severe disabilities preventing mobility;
* Individuals unable to understand or complete the study questionnaire

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will specifically target residents of the Central Division of Fiji, which accounts for approximately 42.7% of Fiji's total population. Most inhabitants are located within the Nausori-Lami corridor, a region characterized by a mix of urban, peri-urban, and rural areas. The Central Division is also notable for its ethnic diversity, comprising Indigenous iTaukei, Indo-Fijians, and other minority groups, making it representative of Fiji's broader demographic composition.
Sampling Method: Probability Sample
Enrollment: 910 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of herd immunity for arboviruses and respiratory viruses by conducting a seroprevalence survey among households including both children and adults In Central division of Fiji | From enrollment to the end of the first inclusion visit (V1) at month 12
  Proportion of participants with Immunoglobulin type G (IgG) antibodies, detected in blood samples : IgG antibodies specific to a panel of arboviruses (including the four DENV serotypes, ZIKV, CHIKV, Ross River virus [RRV], yellow fever virus [YFV], Japanese encephalitis virus [JEV], West Nile virus [WNV]) and respiratory viruses (including influenza viruses A and B, SARS-CoV-2), as well as any major emerging pathogen (pathogen X) will be detected, using a multiplex microsphere immunoassay (MIA). Additionally, seroneutralisation tests will be performed to detect and quantify neutralising antibodies against the same panel of viruses.
  The IgG and neutralising antibody results for each virus will be combined to determine overall immune response (positive/negative) for the targeted viruses.

SECONDARY OUTCOMES:
Evolution of individual memory immunity for arboviruses and respiratory viruses by performing serological monitoring of the study participants over a period of 38 months | From enrollment to the end of the last visit (V4) at month 38
  Proportion of participants with Immunoglobulin type G (IgG) antibodies, detected in blood samples : IgG antibodies specific to a panel of arboviruses (including each of the four DENV serotypes, ZIKV, CHIKV, RRV, YFV, JEV, WNV) and respiratory viruses (including influenza viruses A and B, SARS-CoV-2), as well as any major emerging pathogen (pathogen X) will be detected, using a MIA to track changes in antibody composition (seroconversion or seroreversion) and levels (increase, decrease, or stability), as well as possible cross-reaction phenomena. Additionally, seroneutralisation tests will be performed to detect and quantify neutralising antibodies against the same panel of viruses.
  The IgG and neutralising antibody results for each virus will be combined to determine overall immune response (positive/negative) for the targeted viruses.
Systematic screening and sequencing of acute infections of the study participants over a period of 38 months | From enrollment to the end of the last visit (V4) at month 38
  Systematic screening of acute infections for participants to a panel of arboviruses (including each of the four DENV serotypes, ZIKV, CHIKV, RRV, YFV, JEV, WNV) and respiratory viruses (including influenza viruses A and B, SARS-CoV-2), as well as any major emerging pathogen (pathogen X). Positive samples will undergo whole-genome sequencing.
  This screening and sequencing will allow identification of the viral strain responsible for each infection.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Wilson, MBBS, PhD-Epidemiology, Principal Investigator — Fiji National University
Locations (1):
- Fiji National University, Suva, Central, Fiji